CLINICAL TRIAL: NCT02917044
Title: Use of a High Density Mapping System to Complete Wide Area Circumferential Ablation of the Pulmonary Veins and Avoid Ostial Segmental Ablation
Acronym: HD-WACA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment issues due to competing studies. Higher than expected PVI on first pass. Sample would have to be increased which was not feasible.
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15HH2466
Record Dates: First submitted 2016-08-05; First posted 2016-09-28 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Standard Care (Active Comparator): The operator will attempt to complete the WACA lesion set using standard techniques. These include ablating any obvious gaps in the lesion set, ablating at the WACA line in a location radial to the earliest PV signal measured by the Orion catheter situated within the PV, and guided by amplitude and dV/dt of signals along the WACA lesion set measured using the mapping catheter. If this fails the operator will resort to OSA as per their usual practice.
  Interventions: Procedure: Atrial Fibrillation Ablation; Device: Catheters used to isolate pulmonary veins
- Group B - Rhythmia mapping (Experimental): The operator will form Rhythmia maps focussing on the region of the WACA line surrounding the non-isolated vein(s) whilst pacing from CS. This will be used as a means of targeting RF ablation to gaps in the WACA line (in addition to use of standard observation of signals as per group A). If this fails then the operator will resort to OSA as per their usual practice.
  Interventions: Device: Catheters used to isolate pulmonary veins; Procedure: Atrial Fibrillation Ablation with HD mapping to isolate PVs; Device: Rhythmia HD mapping

INTERVENTIONS:
Procedure: Atrial Fibrillation Ablation — Procedure involving catheter ablation to produce pulmonary vein isolation. Pulmonary veins are isolated by assessing electrograms circumferentially around the PV using the Orion catheter.
  Arms: Group A - Standard Care
Device: Catheters used to isolate pulmonary veins — Catheters transiently inserted into body via femoral veins in order to produce pulmonary vein isolation. These catheters are the same in each arm and comprise the Orion catheter (Boston Scientific) and the Tacticath (St Jude) which are used to produce pulmonary vein isolation and which are approved for use in standard EP procedures by the relevant authorities (CE marked). It is merely the protocol by which they are used that iffers in the two arms.
Procedure: Atrial Fibrillation Ablation with HD mapping to isolate PVs — Procedure involving catheter ablation to produce pulmonary vein isolation. Pulmonary veins are isolated by use of electroanatomical mapping with the Orion catheter around the sites ablation in order to target points of breakthrough.
  Arms: Group B - Rhythmia mapping
Device: Rhythmia HD mapping — Mapping activation patterns using the Rhythmia system in conjunction with the Orion catheter
  Arms: Group B - Rhythmia mapping

SUMMARY:
This is a prospective, multicentre, randomized single blind, parallel group study to be conducted in the UK (2 sites).Approximately 48 patients will be recruited aiming for 40 eligible for randomization. The study is designed to compare the operator's best attempt at WACA completion with and without Rhythmia guidance

DETAILED DESCRIPTION:
BACKGROUND Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia occurring in 1-2% of the general population. AF can be associated with debilitating symptoms and confers an increased risk of death, stroke, heart failure and hospitalization. As such there is a need for effective therapies for AF. In particularly catheter based therapies, which can limit the need for chronic drug therapy, are becoming more widely accepted.

The development of AF requires both a trigger and susceptible substrate. Ectopic activity originating within the pulmonary veins (PVs) is a widely recognised factor in the genesis of paroxysmal AF, whilst electrical, contractile and structural remodelling of atrial myocardium are each important contributing factors to the arrhythmogenic substrate in AF.

An early strategy in paroxysmal AF (PAF) was to target ectopic triggers coming from the PV via ostial segmental ablation (OSA). Here radiofrequency (RF) ablation was applied close to the PV ostia at sites of early signals, usually until PVs were electrically isolated from the left atrium (LA). This approach resulted in a success rate, with regard to freedom from AF after a single procedure, of 65-90% after 1 year but closer to 50% after 5 years. The recognition of PV stenosis as a complication of RF delivery within a PV, as well as the recognition that initiation sites could be located in the antrum led to a shift in ablation strategy towards wider encirclement of the PVs using wide area circumferential ablation (WACA) using electroanatomical mapping to guide RF delivery. This resulted in improved success rates in a head-to-head comparison with OSA and it is possible that this relates to substrate modification inherent in this approach.

Recurrence of AF remains problematic following ablation. Pulmonary vein reconnection after ablation is thought to contribute to the majority of recurrent episodes of AF in paroxysmal AF. Electrical isolation of the PVs is often not achievable with WACA alone - 95% of patients had residual connections following WACA alone in one study. Most clinicians at this juncture will look for any obvious gaps in the line and ablate if there are early PV signals. If this is unsuccessful then it is often necessary to resort to OSA to achieve PV isolation. In essence a large proportion of PV isolation procedures, which started with a WACA strategy, are in fact a hybrid of WACA and OSA. This both has the potential to increase the complication rate by risking PV stenosis and reducing efficacy through omitting important substrate modification and allowing residual connection of part of the antrum and the LA.

The introduction of Rhythmia, a novel electroanatomical mapping system with the potential to rapidly acquire high density electroanatomical data, may allow an alternative strategy and more efficient targeting of gaps in WACA lines. The pilot data shows that the system is particularly adept in assessing gaps in ablation lines including WACA lines. Mapping and targeting such gaps may hold the key to efficiently completing PV isolation after an initial WACA line is performed.

RATIONALE FOR CURRENT STUDY Research Question: Can ostial segmental ablation be avoided during a wide area circumferential ablation (WACA) by using the Rhythmia high density mapping system? Hypothesis: The current study is designed to test the hypothesis that high density mapping using Rhythmia can enhance the operator's ability to electrically isolate PVs without unnecessary excessive ablation or OSA

ELIGIBILITY:
Inclusion Criteria:

* ECG documented AF
* Listed for AF ablation by referring physician
* Planned ablation includes a first-time PVI.
* Patient signed informed consent form

Exclusion Criteria:

* Age <18 or >80
* LA diameter >60mm
* AF secondary to transient correctible abnormalits (e.g. electrolyte imbalance, thyrotoxicosis, recent infective or inflammatory process)
* Intra-atrial thrombus or tumour
* Renal failure requiring haemodialysis
* Heart failure with NYHA III-IV or EF<35%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Total time in minutes required to produce isolation of veins per WACA | Procedural - i.e. assessed over procedure duration only (about 3 hours)
  Following first pass ablation with WACA, if either vein is not isolated the patient will be randomized into group A or B. The total RF time taken to isolate the veins for that WACA will be measured as one of 2 joint primary outcome measures.
Total number of radiofrequency ablation lesions to produce isolation of veins per WACA | Procedural - i.e. assessed over procedure duration only (about 3 hours)
  Following first pass ablation with WACA, if either vein is not isolated the patient will be randomized into group A or B. The total number of lesions (each lesion being 30s in duration) to isolate the veins for that WACA will be measured as one of two joint primary outcome measures.

SECONDARY OUTCOMES:
Whether ostial ablation is required in each case (Yes/No) | Procedural - i.e. assessed over procedure duration only (about 3 hours)
  This is a measure of whether ostial ablation (undesirable) will be required (yes/no). It is assessed during procedure.
Number of radiofrequency ablation lesions required within the WACA lesion set | Procedural - i.e. assessed over procedure duration only (about 3 hours)
  The number of oostial lesions required in each case (number of ablation lesions)
Total radiofrequency ablation time (in mins) within the WACA lesion set | Procedural - i.e. assessed over procedure duration only (about 3 hours)
  This is the total ablation time (in mins) within the WACA required to produce PV isolation
Total number of radiofrequency ablation lesions required to produce PV isolation per patient | Procedural - i.e. assessed over procedure duration only (about 3 hours)
  As per primary endpoint but on a per patient rather than per vein basis
Total procedural time (in mins) required to produce PV isolation | Procedural - i.e. assessed over procedure duration only (about 3 hours)
  Whether procedure time (in mins) is different in group A vs group B
Percentage of patients with successful PV isolation | Procedural - i.e. assessed over procedure duration only (about 3 hours)
  Proportion of veins successfully isolated with the contrasting techniques
Percentage of patients suffering symptomatic PV stenosis | 3 months
  Proportion of patients coming back within 3 months with symptomatic PV stenosis
Percentage of patients with AF recurrence | 3 months
  Proportion of patients remaining AF free at 3 months as analysed per Kaplan-Meier format

CONTACTS AND LOCATIONS:
Overall Officials: Boon Lim, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Hospital, London, Please Select Region, State Or Province, United Kingdom

IPD SHARING:
Plan to Share IPD: No